CLINICAL TRIAL: NCT07179614
Title: Kentucky Women's Justice Community Overdose Innovation Network - Phase II
Acronym: WJCOIN-II
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michele Staton (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Michele Staton, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 106365; RM1DA064496 (NIH)
Record Dates: First submitted 2025-09-16; First posted 2025-09-18 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Overdose Risk; Opioid Use Disorder; Stimulant Use Disorders
Keywords: Overdose; women; criminal justice; opioid use disorder; stimulant use disorder
MeSH Terms: conditions — Opioid-Related Disorders; Drug Overdose

STUDY DESIGN:
Intervention Model Description: 2X2 factorial design includes two levels of pre-release interventions (recovery coaching alone vs. adding support person engagement) and two levels of post-release interventions (prerelease condition alone vs. adding contingency management).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Recovery Coaching Only (Experimental): Following the clinical assessment, all participants will receive the "base" recovery coaching intervention pre-release. RCs will be employed by VOH and will be women with lived experience with OUD/StUD recovery and CLS involvement who will provide strengths-based, person-centered recovery coaching sessions designed to reduce overdose risk. Women will meet with the RC pre-release to assess basic re-entry needs associated with entering treatment (e.g., lack of housing, food, clothing, transportation, employment). RCs will have access to a "barrier relief fund" to address these needs (e.g., clothes for an interview, transportation vouchers) following established RC protocols. At discharge, all women will be provided re-entry transition kits (e.g., hygiene items, condoms, overdose prevention resources) and naloxone.
  Interventions: Behavioral: Overdose Prevention Intervention Package (OPIP)
- Recovery Coaching + Safe Person Engagement (Experimental): Women in this condition will receive the base (RC) pre-release intervention and the Support Person Engagement (SPE) component pre- and post-release. Support Person (SP) designation will draw upon 1) the woman's suggested SP at screening, 2) baseline social network data, and 3) the initial RC meeting. Identified SPs will be screened for eligibility, including being over the age of 18 and willing to engage in intervention sessions. Exclusion criteria for SPs (based on participant and SP self-report) includes past felony conviction, currently incarcerated, on community supervision, or prior history of domestic violence/EPOs. All SPE sessions will align with overdose risk education, understanding treatment options (including MOUD), naloxone distribution, and harm reduction strategies to keep the woman safe during community re-entry. SPs will have access to free naloxone to carry and distribute.
  Interventions: Behavioral: Overdose Prevention Intervention Package (OPIP)
- Recovery Coaching + Contingency Management (Experimental): Women randomized to this group will receive the base pre-release RC intervention, 12 weeks of RC meetings post-release, and 12 weeks of CM post-release. Women will be informed before jail release of the expectations in the CM protocol, target behaviors, and incentive opportunities. The WJCOIN-II CM protocol will be an adapted version of Petry and Martin's approach to reinforce three target verifiable behaviors: 1) meeting with the RC; 2) stimulant abstinence; and 3) opioid abstinence using saliva drug screens. At the conclusion of weekly post-release RC sessions, research staff will join the video call for CM. Virtual CM is feasible, acceptable, and comparable to in-person CM, and research staff will administer CM separately to maintain the integrity of the RC/participant rapport. If the participant does not meet with their RC by the last day of a given week, research staff will contact the participant separately for a CM session.
  Interventions: Behavioral: Overdose Prevention Intervention Package (OPIP)
- Recovery Coaching + Support Person Eng + Contingency Management (Experimental): Women in this intervention condition will participate in the RC condition (pre- and post-release), the SPE sessions (pre- and post-release), and CM post-release.
  Interventions: Behavioral: Overdose Prevention Intervention Package (OPIP)

INTERVENTIONS:
Behavioral: Overdose Prevention Intervention Package (OPIP) — WJCOIN-II's multi-level 2 X 2 randomized factorial design will examine the effectiveness of OPIP components across four study conditions randomly assigned after baseline data collection (n=75 per condition, 100 per jail site), summarized in Table 7 and described below. In addition to group assignment, outcomes will be assessed as a function of engagement in each intervention component defined as the number of sessions attended (RC and CM conditions) and perceived support, which is a count of the number of types of support provided by the RC and SP (e.g., emotional, financial, etc.).

SUMMARY:
This project continues our work with women in the Kentucky Women's Justice Community Overdose Innovation Network Phase II (WJCOIN-II) with the overall aim of reducing overdose risk during the transition from jail to rural communities. WJCOIN-II has potential for significant impact regarding the effectiveness, implementation, and sustainability of innovative overdose prevention strategies during the high-risk time of community re-entry among vulnerable, CLS-involved women in rural communities. This research will impact the field by increasing the capacity of the criminal legal system to respond to the overdose crisis through increased access to prevention strategies to reduce overdose risk.

DETAILED DESCRIPTION:
Overdose deaths among women rose nearly 500% in the past two decades, a rate considerably higher than men. Yet, overdose prevention approaches that target the unique risks of women, particularly those involved in the criminal legal system (CLS) in underserved rural areas, are limited. This application proposes to continue our work with women in the Kentucky Women's Justice Community Overdose Innovation Network Phase II (WJCOIN-II) with the overall aim of reducing overdose risk during the transition from jail to rural communities. Specific aims include: Aim 1: Compare the effectiveness of pre-release RC to RC+SPE in decreasing women's overdose risk during re-entry to rural communities. Through a multi-site 2 X 2 factorial design, women will be randomly assigned to two pre-release conditions (1) Recovery Coaching (RC) only or (2) RC + support person engagement (SPE) to reduce overdose risk through the development of an overdose prevention plan and increase motivation for treatment entry within one-month post-release. Aim 2: Compare the additive effectiveness of CM initiated post-release to RC alone and RC+SPE in decreasing overdose risk and increasing treatment entry and retention among women during re-entry to rural communities. The 2 X 2 factorial randomized design also includes assignment to one of two post-release conditions: 1) continuation of pre-release intervention (RC or RC+SPE) only in the community through ongoing sessions, or 2) addition of contingency management (RC+CM or RC+SPE+CM) to incentivize target behaviors (reduced days of drug use). Depending on treatment entry by the one-month post-release period (non-initiators vs. initiators of treatment), the following aims will be examined post-release from jail: Aim 2a. Among non-initiators, examine the additive effectiveness of post-release CM to reduce overdose risk. Aim 2b. Among treatment initiators, examine the additive effectiveness of post-release CM to increase treatment retention. Aim 3: Contextualize effectiveness of intervention components by examining the roles of perceived acceptability and appropriateness, and identify barriers and facilitators to intervention implementation across the re-entry continuum. Acceptability and appropriateness of intervention components from the perspectives of women and public safety/public health stakeholders (e.g., jail staff, RCs, treatment providers) will be measured through individual-level survey data collection. Aim 4: Examine economic impact of the WJCOIN-II interventions pre-release and post-release in reducing women's overdose risk in rural communities. Cost effectiveness and net societal costs will be assessed by incorporating clinical (overdose risk) and service utilization (treatment entry) outcomes using tailored budget impact tools. The study will make a significant impact regarding the effectiveness, implementation, and sustainability of innovative overdose prevention strategies during the high-risk time of community re-entry among vulnerable, CLS-involved women in rural communities.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 scores of 2+ for opioids (OUD) and/or stimulants (StUD),
* no evidence of cognitive impairment in providing consent,
* a release date within 7-60 days to allow for time for intervention sessions,
* willingness to consider SUD treatment post-release, and
* willingness to provide the name and contact information of at least one person in the community who will support the woman's recovery pre/post-release (SP).

Exclusion Criteria:

* Not living in a rural area
* Any condition that would not allow capable informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-10 (Estimated); Study Completion 2030-10-30 (Estimated)

PRIMARY OUTCOMES:
Overdose risk | 3, 6, and 12 months post-release
  Overdose risk score based on days of opioid, stimulant, and polysubstance use
Treatment entry | 1 month postrelease
  Entry into any formal ASAM level of SUD treatment (e.g., outpatient, intensive outpatient, residential, inpatient, MOUD) (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Staton, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
Pending approval by the IRB and NIDA cooperative

REFERENCES:
- See also: NIH Reporter — https://reporter.nih.gov/